CLINICAL TRIAL: NCT04898348
Title: A Multicenter, Double-blind, Randomized, Placebo-controlled Study to Evaluate the Efficacy and Safety of KBL697 in Patients With Mild to Moderate Active Ulcerative Colitis
Brief Title: A Study to Investigate Efficacy and Safety of KBL697 in Patients With Mild to Moderate Active Ulcerative Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients recruited
Sponsor: KoBioLabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBL-CURE-2020-03
Record Dates: First submitted 2021-05-13; First posted 2021-05-24 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2022-09

CONDITIONS: Ulcerative Colitis
Keywords: microbiome; KBL697; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 3 capsules twice a day dosing of Placebo
  Interventions: Drug: Placebo
- KBL697 (Experimental): 3 capsules twice a day dosing of KBL697
  Interventions: Drug: KBL697

INTERVENTIONS:
Drug: KBL697 — 3 capsules twice a day dosing of KBL697
  Arms: KBL697
Drug: Placebo — 3 capsules twice a day dosing of Placebo
  Arms: Placebo

SUMMARY:
The study is designed to investigate efficacy and safety of KBL697 in patients with mild to moderate active ulcerative colitis. KBL697 has been developed as a potential new treatment for ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Patient has an established diagnosis of ulcerative colitis for at least 3 months prior to Screening
* Patient has active mild to moderate ulcerative colitis at Visit 2
* Patient is taking at least one of the following oral medication: 5-ASA, Corticosteroids, Immunomodulators

Exclusion Criteria:

* Patient has a possible or confirmed diagnosis of Crohn's Disease or other forms of inflammatory bowel disorders
* Patient has a persistent fever of ≥ 38.3°C
* Patient has current signs or symptoms of infection
* Patient has any immunosuppressant condition
* Patient has a known malignancy within 5 years prior to Screening
* Patient who has a medical history of drug abuse or alcohol abuse
* Patient who, in the opinion of the Investigator, has a clinically significant co-morbid disease
* Patient has hepatic failure
* Patient is pregnant or plans a pregnancy within the study period
* Patient has no previous history of treatment for ulcerative colitis (treatment-naïve patient)
* Patient has ongoing or failed treatment for ulcerative colitis with calcineurin inhibitor
* Patient has received biologic medication
* Patient has received antibiotics within 4 weeks prior to Visit 2
* Patient is unable to stop previous antibiotics treatment during study period
* Patient has received probiotics within 2 weeks prior to Visit 2
* Patient with history of major surgery in any region of the gastrointestinal tract
* Patient has received any investigational product or participated in another clinical trial
* Patient has a stool culture or other examination positive for an enteric pathogen
* Patient tests positive for CMV by PCR test at Screening
* Patient tests positive for HIV at Screening
* Exclusion criteria based on results of Hepatitis B at Screening
* Exclusion criteria based on results of Hepatitis C at Screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients with Clinical Remission | Week 8
  Proportion of Patients with Clinical Remission at Week 8

SECONDARY OUTCOMES:
Change from baseline in Partial Mayo Score | Week 8
  Change from baseline in Partial Mayo Score at Week 8 Minimum value: 0, Maximum value: 9, higher score mean a worse outcome
Portion of patients with Endoscopic subscore change | Week 8
  Portion of patients with endoscopic subscore decrease to ≥ 1 at Week 8
Change from baseline in C-reactive Protein | Week 8
  Change from baseline in concentration of C-reactive Protein
Change from baseline in Fecal Calprotectin | Week 8
  Change from baseline in concentration of fecal Calprotectin
Changes from baseline in Inflammatory Bowel Disease Questionnaire score | Week 8
  Changes from baseline in Inflammatory Bowel Disease Questionnaire score Minimum value: 0, Maximum value: 224, higher score mean a worse outcome
Change from baseline in Histologic Disease Activity | Week 8
  Change from baseline in histologic disease activity measured by Geboes score
Safety measure through incidence of treatment-emergent adverse events (TEAEs) | Week 12
  Occurrence of TEAEs, treatment-related TEAEs, TEAEs by severity (mild/moderate/severe), serious TEAEs, TEAEs leading to dose adjustment, treatment termination, or death will be summarized by actual treatment groups respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No